CLINICAL TRIAL: NCT04657887
Title: Observational Registry of Patients With Von WilLEbrand Disease Treated With Voncento®
Brief Title: Registry of Patients With Von WilLEbrand Disease Treated With Voncento®
Acronym: OPALE
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: OPALE study
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Von Willebrand Disease
Keywords: vWD; von Willebrand Factor; vWF
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Voncento® — Solution for injection
  Other Names: Biostate

SUMMARY:
Description of the long-term evolution of patients with von Willebrand disease and treated with Voncento® and of the hemostatic efficacy in the prevention and the treatment of non-surgical bleeding episodes and prevention of surgical bleeding during 2 years after patient inclusion.

DETAILED DESCRIPTION:
Inherited von Willebrand disease (VWD) is considered the most common bleeding disorder. Its prevalence is approximately 1% in the general population but symptomatic patients are rarer (0.01%). It is caused by a partial or total quantitative deficiency (type 1 and type 3) or by a qualitative defect (type 2) of von Willebrand factor (VWF), a large multimeric protein that is required for platelet adhesion and serves as factor VIII (FVIII) carrier. Type 2 VWD is further divided in four subgroups (2A, 2B, 2M, and 2N) that are distinguished according to the nature of the VWF defect. Most patients with type 1 VWD can be treated with the synthetic vasopressin analogue desmopressin (DDAVP; 2-desamino-8-D-arginine vasopressin), whereas patients with type 3 VWD and most patients with type 2 VWD require concentrates containing VWF. Plasma-derived FVIII concentrates, which were initially developed for the treatment of haemophilia, contain large amounts of VWF and are used in patients for whom DDAVP treatment is deemed ineffective or contraindicated. Voncento® (CSL Behring) is a plasma-derived FVIII/VWF concentrate registered in France since 2015 for the treatment and prevention of bleeding events in patients with inherited VWD. OPALE is an observational study describing the use of human coagulation FVIII/VWF concentrate (Voncento®) to treat and prevent bleeding episodes in a French cohort of patients with inherited von Willebrand disease in the real life settings. The aim of the OPALE study is to describe the efficacy and the safety of Voncento® in the prophylaxis and treatment of haemorrhage or surgical bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from constitutional von Willebrand disease for whom Desmopressin treatment is deemed ineffective or contraindicated
* Patients suffering from von Willebrand disease and being treated or having been treated with Voncento® for the treatment of surgical and non-surgical bleeding episodes, the prophylaxis of surgical and non-surgical bleedings
* Patients with no history or suspicion of inhibitors (judged on previous efficacy)

Exclusion Criteria:

* Refusal of the patient or the patient's legal representative to take part in the study;
* Existence of a contraindication to the use of Voncento® treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: French cohort of patients with inherited von Willebrand disease treated with Voncento.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Global assessment by the patient and the investigator of the hemostatic efficacy of Voncento® in the management of non-surgical bleeding episodes | Up to 24 months
Number of non-surgical bleeding episodes per year | Up to 24 months
Number of administrations of Voncento® needed to treat a non-surgical bleeding episode and for the long term prophylaxis | Up to 24 months
Total dose of Voncento® (in IU/kg of VWF) needed to treat a non-surgical bleeding episode and for the long term prophylaxis | Up to 24 months

SECONDARY OUTCOMES:
Assessment by the investigator of the hemostatic efficacy of Voncento® during the treatment and the prophylaxis of surgical bleedings and after surgical procedures | Up to 24 months
Number of administrations of Voncento® needed to prevent or treat surgical bleeding episode | Up to 24 months
Total dose of Voncento® (in IU/kg of VWF) needed to prevent or treat surgical bleeding episode | Up to 24 months
Nature and impact of adverse events and in particular serious adverse events, adverse events related to Voncento® | Up to 24 months
Collection of available biological data (ex: FVIII, VWF:Rco, VWF:Ag) | At baseline and up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring SA
Locations (17):
- France (17):
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Morvan Brest, Brest
  - CHU Lyon, Bron
  - CHU Caen, Caen
  - Hôpital Simone Veil, Eaubonne
  - Hôpital Mignot, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint-Eloi, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Lariboisière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg